CLINICAL TRIAL: NCT03020095
Title: Phase 2 Study To Investigate the Efficacy, Safety And Pharmacokinetics Of Ravidasvir In Combination With Ritonavir-boosted Danoprevir And Ribavirin In Treatment-naive Non-cirrhotic Taiwanese Patients Who Have Chronic Hepatitis C Genotype 1
Brief Title: Efficacy and Safety of Ravidasvir + Danoprevir/r 12-week Oral Therapy in Treatment-Naive Non Cirrhotic G1 CHC Taiwan
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ascletis Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Ascletis Pharma Inc (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ASC162001
Record Dates: First submitted 2017-01-05; First posted 2017-01-13 (Estimated); Results first posted 2020-10-22 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2017-01

CONDITIONS: Chronic Hepatitis C
Keywords: Ravidasvir; HCV GT1; SVR12; Danoprevir/r
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — ravidasvir; danoprevir; Ritonavir; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ravidasvir,Danoprevir/r,RBV (Experimental): Participants will receive Ravidasvir 200mg plus Ritonavir boosted Danoprevir 200/200mg,and Ribavirin 1000/1200mg daily for 12 weeks.
  Interventions: Drug: Ravidasvir; Drug: Danoprevir; Drug: Ritonavir; Drug: Ribavirin

INTERVENTIONS:
Drug: Ravidasvir — Ravidasvir 200mg tablet administered orally once daily
  Other Names: Asclevir
Drug: Danoprevir — Danoprevir 100mg tablet administered orally twice daily
  Other Names: Ganovo
Drug: Ritonavir — Ritonavir 100mg tablet administered orally twice daily
Drug: Ribavirin — Ribavirin(RBV)1000/1200 mg/day (bodyweight<75/≥75 kg)administered orally
  Other Names: Ribasphere®

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety and tolerability of Ravidasvir (ASC16) in combination with Ritonavir-boosted Danoprevir(ASC08) and Ribavirin in treatment-naive no-cirrhotic Taiwanese patients who have chronic hepatitis C genotype1.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent
* Chronic HCV infection (≥6 months) , HCV RNA ≥ 1 × 104 IU/mL
* Never received prior-treatment for HCV with interferon, RBV, or other direct-acting or host-targeting antivirals for HCV
* Chronic liver disease consistent with CHC infection without cirrhosis as determined by biopsy obtained within the past calendar 36 months using one of the liver biopsy methods in the protocol (non-cirrhosis is defined as: Metavir score ˂ 4), or as determined by Fibroscan defined as: ˂ 14.6 kPa. Patients who have not obtained a liver biopsy or Fibroscan in the last 3 years will have a study related Fibroscan performed in order to confirm the diagnosis. Liver biopsy will be performed by investigator's judgement
* All male patients with female partners of childbearing potential must use two reliable forms of effective contraception (combined) during treatment and for 6 months following the last dose of ribavirin
* Others as specified in detailed protocol.

Exclusion Criteria:

* Pregnant or lactating women.
* History or presence of decompensated liver disease (history of ascites, hepatic encephalopathy, HCC, or bleeding esophageal varices)
* Presence or history of non-hepatitis C chronic liver disease, including but not limited to, autoimmune hepatitis, α-1-antitrypsin deficiency, C282Y homozygous hemochromatosis, Wilson's disease, drug- or toxin-induced liver disease, alcohol-related liver disease, primary biliary cirrhosis, sclerosing cholangitis, and porphyria cutanea tarda causing liver pathology or requiring phlebotomy
* Positive hepatitis B surface antigen or HIV antibody at screening
* History or presence of liver cirrhosis
* History of severe psychiatric disease, including psychosis and/or depression, who is not able to participate or able to give written informed consent and to comply with the study restrictions
* History of active malignancy within the last 5 years, with the exception of localized or in situ carcinoma (e.g., basal or squamous cell carcinoma of the skin)
* History of severe cardiac disease (e.g., New York Heart Association Functional Class III or IV, myocardial infarction within 6 months, ventricular tachyarrhythmia's requiring ongoing treatment, unstable angina or other unstable, uncontrolled or significant cardiovascular disease within 6 months). Patients with stable coronary artery disease (e.g., 6 months after by-pass surgery, angioplasty with or without stent placement, etc.) as confirmed by a cardiologist will be permitted. In addition, patients with documented or presumed unstable coronary artery disease, cardiovascular disease, or cerebrovascular disease should not be enrolled.
* Any patient with an increased risk for anemia (e.g., thalassemia, sickle cell anemia, or spherocytosis) or for whom anemia would be medically problematic
* History of pre-existing renal disease, patients with a history of nephrolithiasis will be allowed
* Others as specified in detailed protocol.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2015-08; Primary Completion 2016-08 (Actual); Study Completion 2017-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Huoling Tang, PhD, Study Director — Ascletis Pharmaceuticals Co., Ltd.

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ravidasvir,Danoprevir/r,RBV
Started | 38
Completed | 37
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Ravidasvir,Danoprevir/r,RBV
Number analyzed (Participants) | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.6 (12.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 38
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Taiwan | 38

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Sustained Virologic Response (SVR12) 12 Weeks Post-treatment
Description: SVR12, defined as undetectable HCV RNA 12 weeks after the last day of study drug administration.
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Ravidasvir,Danoprevir/r,RBV
Number analyzed (Participants) | 38
Participants | 38

ADVERSE EVENTS:
Arm/Group | Ravidasvir,Danoprevir/r,RBV
All-Cause Mortality (participants affected / at risk) | 0/38
Serious Adverse Events (participants affected / at risk) | 0/38
Other Adverse Events (participants affected / at risk) | 14/38
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ravidasvir,Danoprevir/r,RBV (N=38)
anemia (Blood and lymphatic system disorders) | 10 (10)
Diarrhea (Gastrointestinal disorders) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Ascletis, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

The study has been completed at all study sites for at least 3 years.